CLINICAL TRIAL: NCT04737850
Title: Safety and Efficacy of Hetrombopag in Children and Adolescents With Chronic Primary Immune Thrombocytopenia：a Randomized, Multicenter, Placebo-controlled Trial
Brief Title: Hetrombopag for Pediatric Patients With Chronic Immune Thrombocytopenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-TPO-ITP-III-PED
Record Dates: First submitted 2021-01-17; First posted 2021-02-04 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — hetrombopag

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PartA, open-label (Experimental): Hetrombopag plus standard of care
  Interventions: Drug: Hetrombopag
- PartB, double-blind treatment group (Experimental): Hetrombopag plus standard of care
  Interventions: Drug: Hetrombopag
- Placebo Comparator (Placebo Comparator): Placebo plus standard of care Part B, double-blind treatment group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hetrombopag — Thrombopoietin receptor agonist
  Arms: PartA, open-label; PartB, double-blind treatment group
Drug: Placebo — Placebo with no active pharmaceutical ingredient
  Arms: Placebo Comparator

SUMMARY:
The purpose of this study is to investigate the efficacy, safety of Hetrombopag in children with previously treated chronic immune thrombocytopenia who are between 6 and 17 years of age. This is a 2 part study. In part A, patients will receive Hetrombopag for 8 weeks. In part B, all patients will receive Hetrombopag for 24 weeks.

DETAILED DESCRIPTION:
This is a two-part, double-blind, randomized, placebo-controlled, and open-label Phase III study to investigate the efficacy, safety of Hetrombopag in pediatric patients with previously treated chronic ITP. In Part A, patients will receive Hetrombopag for 8 weeks. After completing Part A, patients will begin Part B, in which they will be randomized to receive Hetrombopag or placebo in a 12 week double-blind, placebo-controlled treatment period, following an open-label 12 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 6 years old and ≤ 17 years old,both sexes.
2. Part A:Confirmed diagnosis of ITP ≥6months; Part B: Confirmed diagnosis of ITP ≥12months;Platelets <30×10^9/L twice in a row,and platelets <30×10^9/L before taking the medicine.
3. Subjects who are refractory or have relapsed after at least one prior ITP therapy.
4. Birth control during and 28 days after the trial.
5. Written informed consent must be obtained from the patient's guardian and accompanying informed assent from the patient (for children over 8 years old).

Exclusion Criteria:

1. No evidence of other causes of thrombocytopenia.
2. Diagnosis as Evans or Wiskott-Aldrich comprehensive.
3. Patients with any prior history of arterial or venous thrombosis, or diagnosis as thrombophilia.
4. Suffering from serious, progressive, uncontrolled kidney, liver, gastrointestinal, endocrine, lung, heart, nervous system, brain, or mental illness.
5. ALT, AST, or ALP> 1.5 x upper limit of normal (ULN), DBLI, or Scr > 1.2 x upper limit of normal (ULN).
6. Active HIV or HCV-Ab positive,HBsAg positive.
7. PT result exceeds normal by more than ±3s, APTT result exceeds normal by more than ±10s
8. Participated in clinical trials of other drugs (received experimental drugs) within 3 months prior to medication.
9. The inestigators determined that other conditions were inappropriate for participation in this clinical trial.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
the main parameters in population PK/PD modeling in Part A | from baseline to Week 2
  Peak Plasma Concentration (Cmax)
the proportion of patients with a platelet count ≥50×10^9/L at week 10. | from baseline to Week 10
  efficacy in part B

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing children's hospital .Capital medical university, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided